CLINICAL TRIAL: NCT05081414
Title: Efficacy of The Program for Teaching Self-Care in Heart Failure (PEAC-IC): a Randomized Controlled Clinical Trial
Brief Title: Efficacy of the PEAC-IC: a Randomized Controlled Clinical Trial
Acronym: PEAC-IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Michele Nakahara Melo, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-01; PE 1118/2019 (Other Grant/Funding Number: CAPES); Process 2020/15834-8 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2021-09-11; First posted 2021-10-18 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: Nursing; Self-Care; Heart-Failre; Health Education; Clinical Trial
MeSH Terms: conditions — Heart Failure; Health Education

STUDY DESIGN:
Intervention Model Description: PEAC-IC encompasses one presential session and five weekly telephone sessions, focusing on the promotion of self-care and a patient book with all information discussed in the presential session and more 2 diaries, one for the daily weight monitoring and other to assess the symptoms and the and another for monitoring symptoms, making decisions about them and the results obtained. The participants in the intervention group in addition to the patient book will also receive a mechanical scale and a liquid control jar to control the edema and water intake, respectively.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Beyond the active comparator, this group will receive the PEAC-IC, as described previously.
  Interventions: Behavioral: Program for Teaching Self-Care in HF (PEAC-IC)
- Control Group (No Intervention): The Control Group will receive the usual care in the health care institution, which consists of guidance during hospital discharge and delivery of a discharge planning form and outpatient follow-up with medical and nursing consultations and exams when indicated.

INTERVENTIONS:
Behavioral: Program for Teaching Self-Care in HF (PEAC-IC) — As described previously
  Arms: Intervention Group

SUMMARY:
A randomized parallel single-center clinical trial, blinded for the evaluation of the outcomes and statistical analysis. The current hypothesis is that PEAC-IC will improve self-care behavior, knowledge about heart failure, health-related quality of life, and the number of hospitalizations and searches for emergency services in the participants with heart failure.

DETAILED DESCRIPTION:
Heart failure (HF) is an insidious chronic syndrome that impacts the quality of life of people affected by it. One of the ways of controlling the progression of the syndrome is self-care, which involves behaviors to maintain health and to monitor and manage the symptoms of the disease. Several studies have shown that when the person with HF has adequate self-care, there is a reduction in the rate of morbidity and mortality, hospital readmissions, and an improvement in the quality of life. Despite the benefits of self-care, it is still deficient among people with HF in Brazil and worldwide. To improve self-care, educational interventions for the development of skills and behaviors must be performed by nurses, due to their role concerning health education. The Programa Educativo para o Autocuidado na Insuficiência Cardíaca - PEAC-IC is an intervention created to promote the achievement of positive results for people with HF. In a pilot study, PEAC-IC was assessed for acceptability and feasibility, with satisfactory preliminary results. Main objective: To compare the effect of the PEAC-IC with the usual care on self-care behavior, on knowledge about heart failure, on health-related quality of life, and on the number of hospitalizations and searches for emergency services due to HF. Method: This is a randomized parallel single-center clinical trial, blinded for the evaluation of the outcomes and statistical analysis. Participants (1. adults and elderly hospitalized for HF, adults and elderly with HF follow in outpatient care) who meet the participation criteria will be randomized in a simple random way between the intervention and control groups. The intervention group will receive the usual care and the PEAC-IC, offered in one face-to-face session and five structured telephone contacts. The control group will receive only the usual care, which consists of guidance during hospital discharge and delivery of a discharge planning form and outpatient follow-up with medical and nursing consultations and exams when indicated. Both groups will have the outcome variables assessed at baseline, in the seventh week, in the third and sixth months after allocation in the trial. This study will be carried out at the Clinical Cardiological Unit with 42 active beds and a cardiomyopathy outpatient clinic that offer a multidisciplinary health care of approximately 70 clinically stable patients with HF of the Instituto Dante Pazzanese de Cardiologia (IDPC), a public teaching hospital specializing in cardiovascular care. The research will be appreciated by the Research Ethics Committee and will only start after a favorable opinion at the University of São Paulo School of Nursing and the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Be regularly enrolled in the outpatient clinic;
2. Having a confirmed diagnosis of HF, regardless of the etiology or having been hospitalized due to clinical mismatch of the syndrome
3. Have clinical conditions that allow to participate in interviews, as assessed by the researcher;
4. Have an active telephone contact;
5. Be able to listen, speak, read and write portuguese, as assessed by the researcher;

Exclusion Criteria:

1. Patients in the postoperative period of cardiac surgery (up to 60 days after the operation or requiring surgical intervention after inclusion in the study) or any surgical intervention that may increase the demands of self-care.
2. Patients proven to be diagnosed with COVID-19
3. Patients in palliative care, according to the evaluation of the institution's health team, at any time of the research, that is, even after inclusion and randomization.
4. Display adequate self-care and confidence in self-care (≥70 points) on the all EAC-IC subscales (SCHFI 6.2 brazilian version).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Self-care behavior | Self-Care of Heart Failure Index v.6.2 will be assessed at the - T1: research participant allocation, T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  Self-care behavior will be assessed by the Brazilian version of the Self-Care of Heart Failure Index v.6.2 (SCHFI), the Self-Care Scale for Patients with Heart Failure, adapted and validated for use in Brazil. This scale consists of 22 items divided into three subscales. The scores for each subscale can range from 0 to 100 points, and scores equal to or greater than 70, in any subscale, reflect adequate self-care.
Change in Knowledge on Heart Failure | Disease Knowledge Questionnaire will be assessed at the - T1: research participant allocation, T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  The "Disease Knowledge Questionnaire will assess knowledge on Heart failure for Patients with Heart Failure", created and validated for use in Brazil. It consists of 19 items: the HF pathophysiology contents, its concept, diagnosis, risk factors, symptoms, lifestyle habits, treatment, medications used, self-care, and physical exercise. For each item, there are four alternatives: one is the correct answer; one is incomplete; one is incorrect and one is "I don't know". According to the total score obtained, can be categorized as excellent (51 to 57 points); good (40 to 50 points); acceptable (29 to 39 points); little knowledge (17 to 28 points) and insufficient knowledge (< 17 points).

SECONDARY OUTCOMES:
Change in quality of Life | Health-related Quality of Life will be assessed at the - T1: research participant allocation, T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  Quality of Life will be asses using the Minnesota Living with Heart Failure Questionnaire, the validated Portuguese version. The instrument consists of 21 items that assess the participants' perception regarding how much the signs and symptoms of HF made it impossible/limited the daily activities or the activities that the participants would like to perform/perform. These items refer to the physical, emotional and socioeconomic aspects that the presence of HF can impact and the answers range from zero to five points (0: nothing; 1: very little to 5: too much). The final score is obtained through the sum of the answers of the 21 items and can range from zero to 105 points, the higher the score, the worse the quality of life and the lower the score, the better quality of life.
Change in search for emergency medical care due to clinical decompensation of Heart Failure | Will be assessed at the - T1: research participant allocation (number of times during the last 12 months), T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  Number of times reported by the participant or family member/caregiver of fearch for emergency medical care due to clinical decompensation of Heart Failure
Change in hospitalization due to clinical decompensation of Heart Failure | Will be assessed at the - T1: research participant allocation (number of times during the last 12 months), T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  Number of times reported by the participant or family member/caregiver of hospitalization due to clinical decompensation of Heart Failure
Change in feeling of Powerlessness | Will be assessed at the - T1: research participant allocation (number of times during the last 12 months), T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  The feeling of powerlessness will be assessed by the Powerlessness assessment tool, created and validated in adults in the process of hospitalization. It consists of 12 items divided into three domains: the ability to perform a behavior, perception of the ability to make decisions and emotional response to control situations. The possibilities of answering the 12 items range from 'never to 'always' scored from 1 to 5. A cutoff score is not provided for interpreting the results. However, the higher the score, the more intense the feeling of impotence. The score obtained through this instrument will be treated as a continuous quantitative variable, for further categorization under the guidance of a statistician.
Change in Depressive symptoms | Will be assessed at the - T1: research participant allocation (number of times during the last 12 months), T2: seven weeks after allocation, 3 months after T2 and 6 months after T2.
  The Depressive symptoms will be assessed by the Depression Scale CES-D (Center for Epidemiologic Studies Depression Scale) which aims to identify depressive mood and a possible vulnerability to depression. This instrument was created by the NIMH - National Institute of Mental Health and consists of 20 items that measure the occurrence of depressive symptoms, such as mood, somatic symptoms, interactions with other people, and motor functioning, from the frequency of symptoms in the last week to interview. The score for the 20 items can range from 0 to 3 and the response options range from rarely or never, a few times, sometimes, almost always, or always. Thus, the total score varies between zero and sixty points. The occurrence of depressive symptoms is considered from a score of ≥ 16 points

CONTACTS AND LOCATIONS:
Overall Officials: Michele Nakahara-Melo, MsC, Principal Investigator — University of Sao Paulo; Diná Monteiro da Cruz, PhD, Study Chair — University of Sao Paulo; Ana Paula da Conceição, PhD, Study Director — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All variables will be collected and transcribed into the Research Electronic Data Capture (REDCap) application, which will be used for data recording, secure storage, database manipulation. All variables collected will be documented as metadata, and the identity of the participants, such as name and initials, which allow any identification, will be removed from the spreadsheets that will be made available in the repositories. The researcher will keep, outside the application, a listing that will allow the participant to be identified, if necessary during the study. The sharing of metadata in the repositories will be subject to the consent of the participants, and such information will be included in the Consent Form.
  The data will be stored in the cloud and a daily backup of the collected data is provided.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The metadata will be available upon request to the responsible researchers as soon as the research is completed for an indefinite time.
  The researchers responsible for the study that generated the database will be able to, independently, use it for secondary analyses, as long as they ensure reference to the primary study.
Access Criteria: Upon request to the responsible researchers.
URL: https://fapesp.br/gestaodedados

REFERENCES:
- [Background] da Conceicao AP, dos Santos MA, dos Santos B, da Cruz Dde A. Self-care in heart failure patients. Rev Lat Am Enfermagem. 2015 Jul-Aug;23(4):578-86. doi: 10.1590/0104-1169.0288.2591. PMID 26444158
- [Background] Carvalho VO, Guimaraes GV, Carrara D, Bacal F, Bocchi EA. Validation of the Portuguese version of the Minnesota Living with Heart Failure Questionnaire. Arq Bras Cardiol. 2009 Jul;93(1):39-44. doi: 10.1590/s0066-782x2009000700008. English, Portuguese, Spanish. PMID 19838469
- [Result] Ruppar TM, Cooper PS, Johnson ED, Riegel B. Self-care interventions for adults with heart failure: A systematic review and meta-analysis protocol. J Adv Nurs. 2019 Mar;75(3):676-682. doi: 10.1111/jan.13903. Epub 2018 Dec 21. PMID 30397943
- [Result] Sevilla-Cazes J, Ahmad FS, Bowles KH, Jaskowiak A, Gallagher T, Goldberg LR, Kangovi S, Alexander M, Riegel B, Barg FK, Kimmel SE. Heart Failure Home Management Challenges and Reasons for Readmission: a Qualitative Study to Understand the Patient's Perspective. J Gen Intern Med. 2018 Oct;33(10):1700-1707. doi: 10.1007/s11606-018-4542-3. Epub 2018 Jul 10. PMID 29992429
- [Result] Jaarsma T, Hill L, Bayes-Genis A, La Rocca HB, Castiello T, Celutkiene J, Marques-Sule E, Plymen CM, Piper SE, Riegel B, Rutten FH, Ben Gal T, Bauersachs J, Coats AJS, Chioncel O, Lopatin Y, Lund LH, Lainscak M, Moura B, Mullens W, Piepoli MF, Rosano G, Seferovic P, Stromberg A. Self-care of heart failure patients: practical management recommendations from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2021 Jan;23(1):157-174. doi: 10.1002/ejhf.2008. Epub 2020 Oct 20. PMID 32945600
- [Result] Jaarsma T, Stromberg A, Ben Gal T, Cameron J, Driscoll A, Duengen HD, Inkrot S, Huang TY, Huyen NN, Kato N, Koberich S, Lupon J, Moser DK, Pulignano G, Rabelo ER, Suwanno J, Thompson DR, Vellone E, Alvaro R, Yu D, Riegel B. Comparison of self-care behaviors of heart failure patients in 15 countries worldwide. Patient Educ Couns. 2013 Jul;92(1):114-20. doi: 10.1016/j.pec.2013.02.017. Epub 2013 Apr 8. PMID 23579040
- [Result] Riegel B, Dickson VV, Faulkner KM. The Situation-Specific Theory of Heart Failure Self-Care: Revised and Updated. J Cardiovasc Nurs. 2016 May-Jun;31(3):226-35. doi: 10.1097/JCN.0000000000000244. PMID 25774844
- [Result] Vellone E, De Maria M, Iovino P, Barbaranelli C, Zeffiro V, Pucciarelli G, Durante A, Alvaro R, Riegel B. The Self-Care of Heart Failure Index version 7.2: Further psychometric testing. Res Nurs Health. 2020 Dec;43(6):640-650. doi: 10.1002/nur.22083. Epub 2020 Nov 3. PMID 33141495